CLINICAL TRIAL: NCT01490190
Title: Contraceptive Vaginal Ring Releasing Etonogestrel and Ethinylestradiol (NuvaRing): Cycle Control, Acceptability and Tolerability Study in Indian Women
Brief Title: Study of the Use of a Contraceptive Vaginal Ring (NuvaRing) in Normal Daily Practice in Indian Women (P07733)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P07733; CTRI/2011/11/002098 (Registry Identifier: CTRI)
Record Dates: First submitted 2011-11-22; First posted 2011-12-12 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2022-02

CONDITIONS: Contraception
MeSH Terms: interventions — Ethinyl Estradiol; NuvaRing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NuvaRing (Experimental)
  Interventions: Drug: Ethinylestradiol + Etonogestrel Vaginal Ring (NuvaRing)

INTERVENTIONS:
Drug: Ethinylestradiol + Etonogestrel Vaginal Ring (NuvaRing) — Three cycles of NuvaRing use, each cycle consisting of etonogestrel 0.120 mg and ethinylestradiol 0.015 mg over a period of 21 days followed by 7 ring-free days.
  Other Names: NuvaRing; SCH 900702

SUMMARY:
This study will collect information on cycle control, acceptability and tolerability of the vaginal contraceptive ring (NuvaRing) as used in normal daily practice by Indian women.

ELIGIBILITY:
Inclusion Criteria:

* Women at risk of pregnancy and seeking contraception

Exclusion Criteria:

Exclusion criteria based on approved prescribing information in India:

* Presence or history of venous thrombosis, with or without pulmonary embolism.
* Presence or history of arterial thrombosis (e.g. cerebrovascular accident, myocardial infarction) or prodromi of a thrombosis (e.g. angina pectoris or

transient ischemic attack).

* Known predisposition for venous or arterial thrombosis, with or without hereditary involvement such as Activated Protein C (APC) resistance, antithrombin-III deficiency, protein C deficiency, protein S deficiency, hyperhomocysteinemia and antiphospholipid antibodies (anticardiolipin antibodies, lupus anticoagulant).
* History of migraine with focal neurological symptoms.
* Diabetes mellitus with vascular involvement.
* The presence of a severe or multiple risk factor(s) for venous or arterial thrombosis (at the discretion of the doctors)
* Pancreatitis or a history thereof if associated with severe hypertriglyceridemia.
* Presence or history of severe hepatic disease as long as liver function values have not returned to normal.
* Presence or history of liver tumors (benign or malignant).
* Known or suspected malignant conditions of the genital organs or the breasts, if sex steroid-influenced.
* Undiagnosed vaginal bleeding.
* Known or suspected pregnancy.
* Hypersensitivity to the active substances or to any of the excipients of NuvaRing.
* Women who are breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2011-12-26 (Actual); Primary Completion 2012-12-05 (Actual); Study Completion 2012-12-05 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NuvaRing: Safety Population: Safety Population, which included all participants who met inclusion and exclusion criteria and who inserted NuvaRing at least once during the study period.
Period: Overall Study
Arm/Group | NuvaRing: Safety Population
Started | 252
Completed | 204
Not Completed | 48
Not completed — Withdrawal by Subject | 9
Not completed — Adverse Event | 17
Not completed — Protocol Violation | 5
Not completed — Lost to Follow-up | 13
Not completed — Relocation | 1
Not completed — Inconvenience | 1
Not completed — Ring expulsion | 2

BASELINE CHARACTERISTICS:
Arm/Group | NuvaRing: Safety Population
Number analyzed (Participants) | 252
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age data were only available for 218 participants.
  Years | 29.5 (5.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 252
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Regular Menstrual Cycles
Description: The number of participants who experienced regular menstrual bleeding patterns throughout the period of NuvaRing use. Bleeding patterns were to be characterized by particpants as regular or irregular.
Time Frame: Up to 84 days (three 28-day cycles)
Population: Per Protocol Population, which included all participants who completed the study as per protocol.
Measure: Number; unit: Participants
Groups:
- NuvaRing: Three cycles of NuvaRing use, each cycle consisting of etonogestrel 0.120 mg and ethinylestradiol 0.015 mg over a period of 21 days followed by 7 ring-free days.
Arm/Group | NuvaRing
Number analyzed (Participants) | 204
Participants
  First cycle: Regular | 192
  First cycle: Irregular | 9
  First cycle: Missing data | 3
  Second cycle: Regular | 199
  Second cycle: Irregular | 4
  Second cycle: Missing data | 1
  Third cycle: Regular | 200
  Third cycle: Irregular | 3
  Third cycle: Missing data | 1

2. Primary Outcome: Average Number of Bleeding Days Per Cycle
Description: Mean duration of menstruation, per day, per cycle, during the study period.
Time Frame: Up to 84 days (three 28-day cycles)
Population: Per Protocol Population, which included all participants who completed the study as per protocol. Of the total Per Protocol Population (N = 204), data for this outcome measure were missing for 3 partcipants in the first cycle, 1 participant in the second cycle, and 1 participant in the third cycle.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NuvaRing
Number analyzed (Participants) | 203
Days
  First cycle (N = 201) | 3.8 (1.24)
  Second cycle (N = 203) | 3.7 (1.13)
  Third cycle (N = 203) | 3.6 (0.98)

3. Primary Outcome: Average Number of Pads Used Per Day, Per Cycle, During Menstruation While Using Ring
Description: Intensity of menstruation, as indicated by the median number of pads used per day by participants during each cycle of NuvaRing use.
Time Frame: Up to 84 days (three 28-day cycles)
Population: as for outcome 2
Measure: Median (Full Range); unit: Pads
Arm/Group | NuvaRing
Number analyzed (Participants) | 203
Pads
  First cycle (N = 201) | 2 [0 to 6]
  Second cycle (N = 203) | 2 [1 to 10]
  Third cycle (N = 203) | 2 [1 to 7]

4. Primary Outcome: Number of Participants With Intermenstrual Bleeding/Spotting
Description: Number of participants who experienced vaginal bleeding, which includes BLEEDING or SPOTTING, at any time during a cycle other than normal menstruation while in the study. Vaginal bleeding that required >=2 pads per day was classified as BLEEDING. Vaginal bleeding that required <=1 pad per day was classified as SPOTTING.
Time Frame: Up to 84 days (three 28-day cycles)
Population: Per Protocol Population, which included all participants who completed the study as per protocol.
Measure: Number; unit: Participants
Arm/Group | NuvaRing
Number analyzed (Participants) | 204
Participants
  First cycle: Total bleeding/spotting | 5
  First cycle: Bleeding | 1
  First cycle: Spotting | 4
  Second cycle: Total bleeding/spotting | 0
  Second cycle: Bleeding | 0
  Second cycle: Spotting | 0
  Third cycle: Total bleeding/spotting | 1
  Third cycle: Bleeding | 0
  Third cycle: Spotting | 1

5. Primary Outcome: Number of Bleeding Days Per Cycle
Description: Intermenstrual vaginal bleeding that required >=2 pads per day was classified as BLEEDING.
Time Frame: Up to 84 days (three 28-day cycles)
Population: One participant in Per Protocol Population who experienced vaginal bleeding was evaluated for duration of bleeding.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NuvaRing
Number analyzed (Participants) | 1
Days
  First cycle | 4 (0)
  Second cycle | 0 (0)
  Third cycle | 0 (0)

6. Primary Outcome: Number of Spotting Days Per Cycle
Description: Intermenstrual vaginal bleeding that required <=1 pad per day was classified as SPOTTING.
Time Frame: Up to 84 days (three 28-day cycles)
Population: Participants in the Per Protocol Population who experienced spotting were evaluated for duration of spotting.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NuvaRing
Number analyzed (Participants) | 5
Days
  First cycle (N = 4) | 5.5 (4.2)
  Second cycle (N = 0) | 0 (0)
  Third cycle (N = 1) | 3 (0)

7. Primary Outcome: Participants' Assessment of Ease of Insertion of Vaginal Ring
Description: Participants were asked to classify their ability to insert the NuvaRing as very easy, easy, neutral, difficult, very difficult, or failed. The number of participants who responded to each category was reported.
Time Frame: Up to 84 days (three 28-day cycles)
Population: Per Protocol Population, which included all participants who completed the study as per protocol.
Measure: Number; unit: Participants
Arm/Group | NuvaRing
Number analyzed (Participants) | 204
Participants
  First cycle: Very easy | 59
  First cycle: Easy | 82
  First cycle: Neutral | 59
  First cycle: Difficult | 4
  First cycle: Very difficult | 0
  First cycle: Failed | 0
  Second cycle: Very easy | 73
  Second cycle: Easy | 105
  Second cycle: Neutral | 20
  Second cycle: Difficult | 6
  Second cycle: Very difficult | 0
  Second cycle: Failed | 0
  Third cycle: Very easy | 78
  Third cycle: Easy | 113
  Third cycle: Neutral | 12
  Third cycle: Difficult | 1
  Third cycle: Very difficult | 0
  Third cycle: Failed | 0

8. Primary Outcome: Participants' Assessment of Ease of Removal of Vaginal Ring
Description: Participants were asked to classify their ability to remove the NuvaRing as very easy, easy, neutral, difficult, very difficult, or failed. The number of participants who responded to each category was reported.
Time Frame: Up to 84 days (three 28-day cycles)
Population: Per Protocol Population, which included all participants who completed the study as per protocol.
Measure: Number; unit: Participants
Arm/Group | NuvaRing
Number analyzed (Participants) | 204
Participants
  First cycle: Very easy | 70
  First cycle: Easy | 128
  First cycle: Neutral | 6
  First cycle: Difficult | 0
  First cycle: Very difficult | 0
  First cycle: Failed | 0
  Second cycle: Very easy | 81
  Second cycle: Easy | 119
  Second cycle: Neutral | 4
  Second cycle: Difficult | 0
  Second cycle: Very difficult | 0
  Second cycle: Failed | 0
  Third cycle: Very easy | 88
  Third cycle: Easy | 113
  Third cycle: Neutral | 2
  Third cycle: Difficult | 1
  Third cycle: Very different | 0
  Third cycle: Failed | 0

9. Primary Outcome: Participants' Assessment of Feeling Vaginal Ring at Any Time
Description: Participants were asked to assess whether they could feel the NuvaRing at any time and to characterize how often as one of the following: never, rarely, occasionally, mostly, or always. The number of participants who responded to each category was reported.
Time Frame: Up to 84 days (three 28-day cycles)
Population: Per Protocol Population, which included all participants who completed the study as per protocol.
Measure: Number; unit: Participants
Arm/Group | NuvaRing
Number analyzed (Participants) | 204
Participants
  First cycle: Never | 87
  First cycle: Rarely | 89
  First cycle: Occasionally | 25
  First cycle: Mostly | 1
  First cycle: Always | 2
  Second cycle: Never | 107
  Second cycle: Rarely | 86
  Second cycle: Occasionally | 8
  Second cycle: Mostly | 2
  Second cycle: Always | 1
  Third cycle: Never | 117
  Third cycle: Rarely | 79
  Third cycle: Occasionally | 5
  Third cycle: Mostly | 3
  Third cycle: Always | 0

10. Primary Outcome: Participants' Assessment of Feeling Vaginal Ring During Intercourse
Description: Participants were asked to assess whether they could feel the NuvaRing during intercourse and to characterize how often as one the following: never, rarely, occasionally, mostly, or always. The number of participants who responded to each category was reported.
Time Frame: Up to 84 days (three 28-day cycles)
Population: Per Protocol Population, which included all participants who completed the study as per protocol.
Measure: Number; unit: Participants
Arm/Group | NuvaRing
Number analyzed (Participants) | 204
Participants
  First cycle: Never | 85
  First cycle: Rarely | 81
  First cycle: Occasionally | 33
  First cycle: Mostly | 3
  First cycle: Always | 2
  Second cycle: Never | 100
  Second cycle: Rarely | 82
  Second cycle: Occasionally | 21
  Second cycle: Mostly | 0
  Second cycle: Always | 1
  Third cycle: Never | 125
  Third cycle: Rarely | 69
  Third cycle: Occasionally | 9
  Third cycle: Mostly | 0
  Third cycle: Always | 1

11. Primary Outcome: Frequency of Partner Feeling Vaginal Ring During Intercourse
Description: Participants were asked if their partners could feel the NuvaRing during intercourse and to characterize their partners' experience as one of the following: never, rarely, occasionally, mostly, or always. The number of participants who responded to each category was reported.
Time Frame: Up to 84 days (three 28-day cycles)
Population: Per Protocol Population, which included all participants who completed the study as per protocol.
Measure: Number; unit: Participants
Arm/Group | NuvaRing
Number analyzed (Participants) | 204
Participants
  First cycle: Never | 88
  First cycle: Rarely | 75
  First cycle: Occasionally | 34
  First cycle: Mostly | 5
  First cycle: Always | 2
  Second cycle: Never | 112
  Second cycle: Rarely | 65
  Second cycle: Occasionally | 23
  Second cycle: Mostly | 3
  Second cycle: Always | 1
  Third cycle: Never | 121
  Third cycle: Rarely | 69
  Third cycle: Occasionally | 10
  Third cycle: Mostly | 3
  Third cycle: Always | 1

12. Primary Outcome: Frequency of Partner Objecting to Vaginal Ring Use
Description: Participants were asked if their partners objected to their using the NuvaRing during intercourse and to characterize the frequency of their partners' objections as one of the following: never, rarely, occasionally, mostly, or always. The number of participants who responded to each category was reported.
Time Frame: Up to 84 days (three 28-day cycles)
Population: Per Protocol Population, which included all participants who completed the study as per protocol.
Measure: Number; unit: Participants
Arm/Group | NuvaRing
Number analyzed (Participants) | 204
Participants
  First cycle: Never | 129
  First cycle: Rarely | 70
  First cycle: Occasionally | 4
  First cycle: Mostly | 1
  First cycle: Always | 0
  Second cycle: Never | 143
  Second cycle: Rarely | 55
  Second cycle: Occasionally | 5
  Second cycle: Mostly | 1
  Second cycle: Always | 0
  Third cycle: Never | 153
  Third cycle: Rarely | 45
  Third cycle: Occasionally | 3
  Third cycle: Mostly | 3
  Third cycle: Always | 0

13. Primary Outcome: Participants' Overall Satisfaction With Vaginal Ring
Description: Participants were asked to characterize their overall satisfaction with the NuvaRing as one of the following: very satisfied, satisfied, neutral, unsatisfied, or very unsatisfied. The number of participants who responded to each category was reported.
Time Frame: Up to 84 days (three 28-day cycles)
Population: Safety Population, which included all participants who met inclusion and exclusion criteria and who inserted NuvaRing at least once during the study period.
Measure: Number; unit: Participants
Arm/Group | NuvaRing
Number analyzed (Participants) | 252
Participants
  First cycle (N = 252): Very satisfied | 68
  First cycle (N = 252): Satisfied | 119
  First cycle (N = 252): Neutral | 28
  First cycle (N = 252): Unsatisfied | 9
  First cycle (N = 252): Very unsatisfied | 1
  First cycle (N = 252): Missing data | 27
  Second cycle (N = 213): Very satisfied | 82
  Second cycle (N = 213): Satisfied | 112
  Second cycle(N = 213): Neutral | 15
  Second cycle (N = 213): Unsatisfied | 1
  Second cycle (N = 213): Very unsatisfied | 0
  Second cycle (N = 213): Missing data | 3
  Third cycle (N = 207): Very satisfied | 88
  Third cycle (N = 207): Satisfied | 107
  Third cycle (N = 207): Neutral | 9
  Third cycle (N = 207): Unsatisfied | 1
  Third cycle (N = 207): Very unsatisfied | 1
  Third cycle (N = 207): Missing data | 1

14. Primary Outcome: Number of Participants Who Plan to Continue Using Vaginal Ring
Description: Participants were asked at follow-up visits after every cycle whether they planned to continue using NuvaRing, and their answers were recorded.
Time Frame: Up to 84 days (three 28-day cycles)
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | NuvaRing
Number analyzed (Participants) | 252
Participants
  First cycle (N = 252): Yes | 216
  First cycle (N = 252): No | 9
  First cycle (N = 252): Missing data | 27
  Second cycle (N = 213): Yes | 205
  Second cycle (N = 213): No | 5
  Second cycle (N = 213): Missing data | 3
  Third cycle (N = 207): Yes | 159
  Third cycle (N = 207): No | 47
  Third cycle (N = 207): Missing data | 1

15. Primary Outcome: Number of Participants Who Would Recommend Vaginal Ring to Others
Description: Participants were asked at follow-up visits after every cycle whether they would recommend NuvaRing to other women, and their answers were reported.
Time Frame: Up to 84 days (three 28-day cycles)
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | NuvaRing
Number analyzed (Participants) | 252
Participants
  First cycle (N = 252): Yes | 208
  First cycle (N = 252): No | 16
  First cycle (N = 252): Missing data | 28
  Second cycle (N = 213): Yes | 197
  Second cycle (N = 213): No | 13
  Second cycle (N = 213): Missing data | 3
  Third cycle (N = 207): Yes | 193
  Third cycle (N = 207): No | 13
  Third cycle (N = 207): Missing data | 1

16. Secondary Outcome: Number of Pregnancies Due to Contraceptive Method Failure During the Study
Description: For participants with suspected pregnancy during in-treatment period, pregnancy was to be confirmed by hCG qualitative analysis using strip and/or other test(s) at the discretion of the treating physician.
Time Frame: Up to 84 days (three 28-day cycles)
Population: as for outcome 13
Measure: Number; unit: Pregnancies
Arm/Group | NuvaRing
Number analyzed (Participants) | 252
Pregnancies
  First cycle (N = 252): Yes | 0
  First cycle (N = 252): No | 226
  First cycle (N = 252): Missing data | 26
  Second cycle (N = 213): Yes | 0
  Second cycle (N = 213): No | 210
  Second cycle (N = 213): Missing data | 3
  Third cycle (N = 207): Yes | 0
  Third cycle (N = 207): No | 207
  Third cycle (N = 207): Missing data | 0

17. Secondary Outcome: Number of Participants Who Reported at Least One Adverse Event During the Study
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product, biologic, or medical device, which does not necessarily have a causal relationship with the treatment.
Time Frame: Up to 84 days (three 28-day cycles)
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | NuvaRing
Number analyzed (Participants) | 252
Participants | 47

18. Secondary Outcome: Number of Participants Who Reported a Serious Adverse Event During the Study
Description: A serious adverse event is any adverse drug or biologic or device experience that results in death, a life-threatening adverse event, persistent or significant disability or incapacity; requires in-patient hospitalization, or prolonged hospitalization; or causes a congenital anomaly or birth defect.
Time Frame: Up to 84 days (three 28-day cycles)
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | NuvaRing
Number analyzed (Participants) | 252
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 84 days (three 28-day cycles)
Arm/Group | NuvaRing: Safety Population
Serious Adverse Events (participants affected / at risk) | 0/252
Other Adverse Events (participants affected / at risk) | 13/252
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NuvaRing: Safety Population (N=252)
Vaginal haemorrhage (Reproductive system and breast disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator agrees not to publish or publicly present interim results of the Study without prior written consent of sponsor, agrees to provide 45 days written notice to sponsor prior to submission for publication or presentation, and permits sponsor to review copies of abstracts and manuscripts for publication, and slides and text of oral presentations and text of any electronically transmitted media such as the Internet, World Wide Web, etc.